CLINICAL TRIAL: NCT04974632
Title: Mobile 3D C-arm CT for Lung Tumor Localization Efficacy Analysis: a Prospective Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202100442A3
Record Dates: First submitted 2021-07-21; First posted 2021-07-23 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2021-07

CONDITIONS: Lung Tumor; Thoracoscopic Surgery
Keywords: Lung tumor; mobile 3D C-arm computed tomography(CT); Video-assisted thoracoscopic surgery (VATS)
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- localization (Other): small, deep or ground-glass opacity (GGO) lung tumor, Mobile 3D C-arm CT assisted pre-operative localization, video-assisted thoracic surgery(VATS)
  Interventions: Procedure: localization

INTERVENTIONS:
Procedure: localization — small, deep or ground-glass opacity (GGO) lung tumor, Mobile 3D C-arm CT assisted pre-operative localization, video-assisted thoracic surgery(VATS)

SUMMARY:
It is well known that video-assisted thoracoscopic surgery (VATS) is preferred to open surgery for lung resection because of the smaller incisions and optimized postoperative recovery, including a shorter length of hospitalization and much decreased local tenderness. Studies have shown less operative and post-operative morbidity with decreased operative times. However, for small nodules (i.e. lesions <1 cm or those at a distance more than 1.5cm from the lung periphery), adequate identiﬁcation of the target nodule has been being difficult by VATS with necessity of more significant resection or thoracotomy conversion to ensure complete tumor resection.

In order to improve nodule localization, a variety of preoperative localization methods such as CT-guide hook wire or methyl blue dye localization have been proposed. It has been proved to be much easier to mark lung nodules and help guide resection during VATS. However, there are certain concerns. First, it is difficult to minimize the time between the localization procedure and the subsequent surgery in reality. Second, there is concern for patient safety, in particular pneumothorax or hemothorax, during transferred to and from the ward to the radiology suit and in the frequent delays and waiting in reception areas prior to transfer to operating theaters. Finally, interdepartmental transfers and delays can also increase the risk of hook wire dislodgement.

Theoretically, the aforementioned disadvantage could be solved by performing the localization procedure and the lung surgery in the same operating room environment. We performed single-step localization and removal of small pulmonary nodules in the hybrid OR equipped with floor-mounted C-arm cone-beam computed tomography (CBCT) in the previous study. However, it costed a lot of money and every localization could only be performed in the hybrid OR. Mobile 3D C-arm CT is another form of CBCT. It depicts soft tissues with high contrast but also offer a more affordable solution with relative low cost. In this case series, we will investigate the use of a mobile 3D C-arm CT for single-step localization and removal of small pulmonary nodules.

DETAILED DESCRIPTION:
Pre-operative CT scans will be used for localization planning. The images will be reviewed by our team to determine optimal placement of wires or indocyanine green. After induction of general anesthesia and insertion of a double-lumen tube, the patient will be placed in either supine, prone or lateral decubitus position. Under end-inspiratory breath-hold, an initial 30 second rotary scan for surgical planning will be obtained. The puncture path will be planned to be as short as possible while avoiding transfissural punctures or being oriented towards major vascular structure. The skin entry site for the planned needle puncture route will then identified under the guidance of the referential metallic marker. An 18-gauze marker needle will be gradually advanced under CT-guidance until it reached the target lesion. A total of 0.3 ml ICG dye(for superficial lesion) or microcoil or hookwire(for deeper lesion) will then be used to localize the tumor.

ELIGIBILITY:
Inclusion Criteria:

<1 cm, those at a distance more than 1.5 cm from the lung periphery, or ground-glass opacity (GGO) lung lesion.

Exclusion Criteria:

Age <20 serious pulmonary heart disease more than one tumors needed localization

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Procedure time | from initiation of the procedure time (first time CT scanning) to the end (localization complete).
  Recording the time of localization procedure, including needle puncture time.
success rate of localization | from initiation of localization to completion of surgery
  Recording the result of localization (success or not), the failure reason, and the deviation distance

SECONDARY OUTCOMES:
Radiation dose | from initiation of the preprocedural CT scanning to the end of the postprocedural CT scanning, through study completion, an average of 1 year.
  Effective dose estimates were performed using thermoluminescent dosimeters (TLD).
Complication rate | from initiation of localization to completion of surgery
  Recording the rate of common complications, such as pneumothorax, hemothorax.

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Kai Chao, MD, Ph D, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang BY, Huang JY, Cheng CY, Lin CH, Ko J, Liaw YP. Lung cancer and prognosis in taiwan: a population-based cancer registry. J Thorac Oncol. 2013 Sep;8(9):1128-35. doi: 10.1097/JTO.0b013e31829ceba4. PMID 23945383
- [Background] Huang HL, Kung PT, Chiu CF, Wang YH, Tsai WC. Factors associated with lung cancer patients refusing treatment and their survival: a national cohort study under a universal health insurance in Taiwan. PLoS One. 2014 Jul 7;9(7):e101731. doi: 10.1371/journal.pone.0101731. eCollection 2014. PMID 24999633
- [Background] Bach PB, Mirkin JN, Oliver TK, Azzoli CG, Berry DA, Brawley OW, Byers T, Colditz GA, Gould MK, Jett JR, Sabichi AL, Smith-Bindman R, Wood DE, Qaseem A, Detterbeck FC. Benefits and harms of CT screening for lung cancer: a systematic review. JAMA. 2012 Jun 13;307(22):2418-29. doi: 10.1001/jama.2012.5521. PMID 22610500
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Oken MM, Hocking WG, Kvale PA, Andriole GL, Buys SS, Church TR, Crawford ED, Fouad MN, Isaacs C, Reding DJ, Weissfeld JL, Yokochi LA, O'Brien B, Ragard LR, Rathmell JM, Riley TL, Wright P, Caparaso N, Hu P, Izmirlian G, Pinsky PF, Prorok PC, Kramer BS, Miller AB, Gohagan JK, Berg CD; PLCO Project Team. Screening by chest radiograph and lung cancer mortality: the Prostate, Lung, Colorectal, and Ovarian (PLCO) randomized trial. JAMA. 2011 Nov 2;306(17):1865-73. doi: 10.1001/jama.2011.1591. Epub 2011 Oct 26. PMID 22031728
- [Background] Humphrey LL, Deffebach M, Pappas M, Baumann C, Artis K, Mitchell JP, Zakher B, Fu R, Slatore CG. Screening for lung cancer with low-dose computed tomography: a systematic review to update the US Preventive services task force recommendation. Ann Intern Med. 2013 Sep 17;159(6):411-420. doi: 10.7326/0003-4819-159-6-201309170-00690. PMID 23897166
- [Background] US Preventive Services Task Force; Krist AH, Davidson KW, Mangione CM, Barry MJ, Cabana M, Caughey AB, Davis EM, Donahue KE, Doubeni CA, Kubik M, Landefeld CS, Li L, Ogedegbe G, Owens DK, Pbert L, Silverstein M, Stevermer J, Tseng CW, Wong JB. Screening for Lung Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2021 Mar 9;325(10):962-970. doi: 10.1001/jama.2021.1117. PMID 33687470
- [Background] Suzuki K, Nagai K, Yoshida J, Ohmatsu H, Takahashi K, Nishimura M, Nishiwaki Y. Video-assisted thoracoscopic surgery for small indeterminate pulmonary nodules: indications for preoperative marking. Chest. 1999 Feb;115(2):563-8. doi: 10.1378/chest.115.2.563. PMID 10027460
- [Background] Santambrogio R, Montorsi M, Bianchi P, Mantovani A, Ghelma F, Mezzetti M. Intraoperative ultrasound during thoracoscopic procedures for solitary pulmonary nodules. Ann Thorac Surg. 1999 Jul;68(1):218-22. doi: 10.1016/s0003-4975(99)00459-2. PMID 10421144
- [Background] Kim YD, Jeong YJ, I H, Cho JS, Lee JW, Kim HJ, Lee SH, Kim DH. Localization of pulmonary nodules with lipiodol prior to thoracoscopic surgery. Acta Radiol. 2011 Feb 1;52(1):64-9. doi: 10.1258/ar.2010.100307. PMID 21498328
- [Background] Mayo JR, Clifton JC, Powell TI, English JC, Evans KG, Yee J, McWilliams AM, Lam SC, Finley RJ. Lung nodules: CT-guided placement of microcoils to direct video-assisted thoracoscopic surgical resection. Radiology. 2009 Feb;250(2):576-85. doi: 10.1148/radiol.2502080442. PMID 19188326
- [Background] Finley RJ, Mayo JR, Grant K, Clifton JC, English J, Leo J, Lam S. Preoperative computed tomography-guided microcoil localization of small peripheral pulmonary nodules: a prospective randomized controlled trial. J Thorac Cardiovasc Surg. 2015 Jan;149(1):26-31. doi: 10.1016/j.jtcvs.2014.08.055. Epub 2014 Sep 16. PMID 25293355
- [Background] Cheng C, Fang HY, Wen CT, Chao YK. Real-time image-guided electromagnetic navigation bronchoscopy dual-marker technique to localize deep pulmonary nodules in a hybrid operating room. Eur J Cardiothorac Surg. 2020 Aug 1;58(Suppl_1):i103-i105. doi: 10.1093/ejcts/ezz360. PMID 32105309
- [Background] Sadoughi A, Virdi S. Mobile 3D Intraprocedural Fluoroscopy in Combination With Ultrathin Bronchoscopy for Biopsy of Peripheral Lung Nodules. J Bronchology Interv Pulmonol. 2021 Jan 1;28(1):76-80. doi: 10.1097/LBR.0000000000000711. PMID 32947357
- [Background] Kpodonu J, Raney A. The cardiovascular hybrid room a key component for hybrid interventions and image guided surgery in the emerging specialty of cardiovascular hybrid surgery. Interact Cardiovasc Thorac Surg. 2009 Oct;9(4):688-92. doi: 10.1510/icvts.2009.209429. Epub 2009 Jul 21. PMID 19622541
- [Background] Biasi L, Ali T, Ratnam LA, Morgan R, Loftus I, Thompson M. Intra-operative DynaCT improves technical success of endovascular repair of abdominal aortic aneurysms. J Vasc Surg. 2009 Feb;49(2):288-95. doi: 10.1016/j.jvs.2008.09.013. Epub 2008 Nov 28. PMID 19038527
- [Background] Heran NS, Song JK, Namba K, Smith W, Niimi Y, Berenstein A. The utility of DynaCT in neuroendovascular procedures. AJNR Am J Neuroradiol. 2006 Feb;27(2):330-2. PMID 16484404
- [Background] Irie K, Murayama Y, Saguchi T, Ishibashi T, Ebara M, Takao H, Abe T. Dynact soft-tissue visualization using an angiographic C-arm system: initial clinical experience in the operating room. Neurosurgery. 2008 Mar;62(3 Suppl 1):266-72; discussion 272. doi: 10.1227/01.neu.0000317403.23713.92. PMID 18424996
- [Background] Fang HY, Chao YK, Hsieh MJ, Wen CT, Ho PH, Tang WJ, Liu YH. Image-guided video-assisted thoracoscopic surgery for small ground glass opacities: a case series. J Vis Surg. 2017 Oct 18;3:142. doi: 10.21037/jovs.2017.09.08. eCollection 2017. PMID 29302418
- [Background] Hsieh MJ, Wen CT, Fang HY, Wen YW, Lin CC, Chao YK. Learning curve of image-guided video-assisted thoracoscopic surgery for small pulmonary nodules: A prospective analysis of 30 initial patients. J Thorac Cardiovasc Surg. 2018 Apr;155(4):1825-1832.e1. doi: 10.1016/j.jtcvs.2017.11.079. Epub 2017 Dec 13. PMID 29338860
- [Background] Chao YK, Wen CT, Fang HY, Hsieh MJ. A single-center experience of 100 image-guided video-assisted thoracoscopic surgery procedures. J Thorac Dis. 2018 Jun;10(Suppl 14):S1624-S1630. doi: 10.21037/jtd.2018.04.44. PMID 30034827
- [Background] Chao YK, Pan KT, Wen CT, Fang HY, Hsieh MJ. A comparison of efficacy and safety of preoperative versus intraoperative computed tomography-guided thoracoscopic lung resection. J Thorac Cardiovasc Surg. 2018 Nov;156(5):1974-1983.e1. doi: 10.1016/j.jtcvs.2018.06.088. Epub 2018 Jul 20. PMID 30119900
- [Background] Fang HY, Chang KW, Chao YK. Hybrid operating room for the intraoperative CT-guided localization of pulmonary nodules. Ann Transl Med. 2019 Jan;7(2):34. doi: 10.21037/atm.2018.12.48. PMID 30854387
- [Background] Gill RR, Zheng Y, Barlow JS, Jayender J, Girard EE, Hartigan PM, Chirieac LR, Belle-King CJ, Murray K, Sears C, Wee JO, Jaklitsch MT, Colson YL, Bueno R. Image-guided video assisted thoracoscopic surgery (iVATS) - phase I-II clinical trial. J Surg Oncol. 2015 Jul;112(1):18-25. doi: 10.1002/jso.23941. Epub 2015 May 28. PMID 26031893
- [Background] Ng CSH, Man Chu C, Kwok MWT, Yim APC, Wong RHL. Hybrid DynaCT scan-guided localization single-port lobectomy. [corrected]. Chest. 2015 Mar;147(3):e76-e78. doi: 10.1378/chest.14-1503. PMID 25732474
- [Background] Rouze S, de Latour B, Flecher E, Guihaire J, Castro M, Corre R, Haigron P, Verhoye JP. Small pulmonary nodule localization with cone beam computed tomography during video-assisted thoracic surgery: a feasibility study. Interact Cardiovasc Thorac Surg. 2016 Jun;22(6):705-11. doi: 10.1093/icvts/ivw029. Epub 2016 Feb 26. PMID 26921886
- [Derived] Fang HY, Cheng C, Chou PL, Chao YK. Feasibility and Efficacy of Mobile Three-Dimensional c-Arm Systems for Single-Stage Localization and Resection of Small Pulmonary Nodules: A Pilot Clinical Trial. Interdiscip Cardiovasc Thorac Surg. 2026 Jan 6;41(1):ivaf313. doi: 10.1093/icvts/ivaf313. PMID 41428415